CLINICAL TRIAL: NCT00835627
Title: Medication and Psychotherapy Treatment Trial for Psychogenic Nonepileptic Seizures
Brief Title: Treatment Trial for Psychogenic Nonepileptic Seizures
Acronym: NEST-T_1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: American Epilepsy Society (Other); Epilepsy Foundation (Other); University of Cincinnati (Other); Stanford University (Other)
Responsible Party: Principal Investigator, W. Curt LaFrance Jr., M.D., Director, Neuropsychiatry and Behavioral Neurology, Rhode Island Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EF122982
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Convulsion, Non-Epileptic; Conversion Disorder; Depression; Stress Disorders, Post-Traumatic; Dissociative Disorders
Keywords: Treatment; Cognitive Behavior Therapy; pharmacotherapy; psychogenic nonepileptic seizures; pseudoseizures; dissociative seizures; conversion disorder
MeSH Terms: conditions — Seizures; Conversion Disorder; Depression; Stress Disorders, Post-Traumatic; Dissociative Disorders; Psychogenic Nonepileptic Seizures | interventions — Sertraline; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- sertraline (Active Comparator): flexible dose sertraline
  Interventions: Drug: sertraline
- CBT-ip (Active Comparator): cognitive behavioral therapy-informed psychotherapy for nonepileptic seizures: 12 individual, 1 hour therapy sessions
  Interventions: Behavioral: CBT-ip
- Combined (sertraline + CBT-ip) (Active Comparator): flexible dose sertraline and cognitive behavioral therapy-informed psychotherapy for nonepileptic seizures: flexible dose sertraline and 12 individual, 1 hour therapy sessions
  Interventions: Other: Combined (sertraline + CBT-ip)
- Standard care (Active Comparator): community care / treatment as usual: routine follow up with existing providers
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: sertraline — flexible dose sertraline
  Other Names: Zoloft
  Arms: sertraline
Behavioral: CBT-ip — cognitive behavioral therapy-informed psychotherapy for nonepileptic seizures: 12 individual 1 hour therapy sessions
  Arms: CBT-ip
Other: Combined (sertraline + CBT-ip) — flexible dose sertraline and cognitive behavioral therapy-informed psychotherapy for nonepileptic seizures: flexible dose sertraline and 12, individual 1 hour therapy sessions
  Other Names: Zoloft; CBT-ip
  Arms: Combined (sertraline + CBT-ip)
Other: Standard Care — community care, treatment as usual: routine follow up with existing providers
  Other Names: TAU, standard care
  Arms: Standard care

SUMMARY:
The investigators propose that patients who receive targeted pharmacotherapy (sertraline) or focused psychotherapy (cognitive behavioral therapy-informed psychotherapy (CBT-ip) for NES) or combined treatment (CBT-ip + sertraline) will report fewer nonepileptic seizures (NES) compared to patients who receive community care / treatment as usual (TAU). The purpose of this study is to provide pilot testing and data to inform the future multicenter randomized controlled trial based on the hypothesis.

DETAILED DESCRIPTION:
This is a pilot, prospective, multi-center, randomized controlled trial, that assesses the number of NES in patients treated with either flexible dose sertraline (Zoloft), cognitive behavioral therapy-informed psychotherapy (CBT-ip), combined therapy (sertraline + CBT-ip) or community care (treatment as usual TAU). This study will provide outcomes data and the effect size necessary for a future R01, multi-center randomized control trial. Secondary objective variables include reduction in depression, anxiety, impulsivity scores, and improvement in psychosocial functioning.

After being diagnosed with NES by video EEG monitoring (vEEG), up to 40 participants will be enrolled and monitored during a two week lead in period for their baseline NES and psychosocial symptoms and functioning. At week 2, they will be randomized to either: flexible dose sertraline (25 to 200mg), CBT, CBT+med, or to the control arm, TAU. Participants randomized to the sertraline arm will be titrated over 6 weeks up to 200mg or to dose limited by side effects. The subjects will stay on their maximum fixed dose for the next 4 weeks. At week 10, the subjects may elect to remain on the sertraline or they can taper off the medication over the final two weeks of the treatment trial. Those randomized to the CBT-ip arm will receive 12 weekly sessions of CBT-ip for NES. Those randomized to the CBT-ip + med arm will receive both treatments. Those randomized to the TAU arm will follow with their treatment providers.

After the treatment trial, the subjects will have follow up phone calls at month 4, 8, and 12 after enrollment to assess seizure status, medication usage, and global functioning.

Upon enrollment, subjects will be evaluated with a structured psychiatric and neurological exam, and with bi-weekly, 30 to 60 minute appointments where they will complete symptom and function scales. They will keep a seizure diary to evaluate their daily seizure activity.

ELIGIBILITY:
Inclusion Criteria:

* Video electroencephalogram (EEG) confirmed diagnosis of NES
* Have at least one nonepileptic seizure per month
* Able to complete self report symptom scales
* Not receiving optimized sertraline

Exclusion Criteria:

* Equivocal EEG findings
* using monoamine oxidase inhibitors (MAOIs), pimozide, or sumatriptan
* allergy/sensitivity to sertraline
* current alcohol/drug dependence
* serious medical illness requiring current hospitalization

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
seizure frequency | weekly

SECONDARY OUTCOMES:
Identify predictors of response from the following 3 groups: clinical diagnoses | baseline
psychological symptoms | bi-weekly
socio-demographic variables | bi-weekly

CONTACTS AND LOCATIONS:
Overall Officials: W. Curt LaFrance, Jr., MD, MPH, Principal Investigator — Rhode Island Hospital / Brown Medical School
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - University of Cincinnati, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Background] LaFrance WC. How many patients with psychogenic nonepileptic seizures also have epilepsy? Neurology. 2002 Mar 26;58(6):990; author reply 990-1. doi: 10.1212/wnl.58.6.990. No abstract available. PMID 11914432
- [Background] LaFrance WC Jr, Devinsky O. Treatment of nonepileptic seizures. Epilepsy Behav. 2002 Oct;3(5 Suppl):19-23. doi: 10.1016/s1525-5069(02)00505-4. PMID 12609316
- [Background] LaFrance WC Jr, Devinsky O. The treatment of nonepileptic seizures: historical perspectives and future directions. Epilepsia. 2004;45 Suppl 2:15-21. doi: 10.1111/j.0013-9580.2004.452002.x. PMID 15186340
- [Background] LaFrance WC Jr, Barry JJ. Update on treatments of psychological nonepileptic seizures. Epilepsy Behav. 2005 Nov;7(3):364-74. doi: 10.1016/j.yebeh.2005.07.010. Epub 2005 Sep 16. PMID 16150653
- [Background] LaFrance WC Jr, Alper K, Babcock D, Barry JJ, Benbadis S, Caplan R, Gates J, Jacobs M, Kanner A, Martin R, Rundhaugen L, Stewart R, Vert C; NES Treatment Workshop participants. Nonepileptic seizures treatment workshop summary. Epilepsy Behav. 2006 May;8(3):451-61. doi: 10.1016/j.yebeh.2006.02.004. Epub 2006 Mar 15. PMID 16540377
- [Background] LaFrance WC Jr. Use of serum prolactin in diagnosing epileptic seizures: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2006 Apr 25;66(8):1287-8; author reply 1287-8. doi: 10.1212/01.wnl.0000222496.94195.14. No abstract available. PMID 16636265
- [Background] LaFrance WC Jr, Benbadis SR. Avoiding the costs of unrecognized psychological nonepileptic seizures. Neurology. 2006 Jun 13;66(11):1620-1. doi: 10.1212/01.wnl.0000224953.94807.be. No abstract available. PMID 16769930
- [Background] LaFrance WC Jr, Blum AS, Miller IW, Ryan CE, Keitner GI. Methodological issues in conducting treatment trials for psychological nonepileptic seizures. J Neuropsychiatry Clin Neurosci. 2007 Fall;19(4):391-8. doi: 10.1176/jnp.2007.19.4.391. PMID 18070841
- [Background] LaFrance WC Jr, Rusch MD, Machan JT. What is "treatment as usual" for nonepileptic seizures? Epilepsy Behav. 2008 Apr;12(3):388-94. doi: 10.1016/j.yebeh.2007.12.017. Epub 2008 Feb 20. PMID 18282812
- [Background] LaFrance WC Jr. Psychogenic nonepileptic seizures. Curr Opin Neurol. 2008 Apr;21(2):195-201. doi: 10.1097/WCO.0b013e3282f7008f. PMID 18317280
- [Background] LaFrance WC Jr, Baker GA, Duncan R, Goldstein LH, Reuber M. Minimum requirements for the diagnosis of psychogenic nonepileptic seizures: a staged approach: a report from the International League Against Epilepsy Nonepileptic Seizures Task Force. Epilepsia. 2013 Nov;54(11):2005-18. doi: 10.1111/epi.12356. Epub 2013 Sep 20. PMID 24111933
- [Background] LaFrance WC Jr, Reuber M, Goldstein LH. Management of psychogenic nonepileptic seizures. Epilepsia. 2013 Mar;54 Suppl 1:53-67. doi: 10.1111/epi.12106. PMID 23458467
- [Background] LaFrance WC Jr, Deluca M, Machan JT, Fava JL. Traumatic brain injury and psychogenic nonepileptic seizures yield worse outcomes. Epilepsia. 2013 Apr;54(4):718-25. doi: 10.1111/epi.12053. Epub 2013 Jan 2. PMID 23281644
- [Background] LaFrance WC Jr, Alosco ML, Davis JD, Tremont G, Ryan CE, Keitner GI, Miller IW, Blum AS. Impact of family functioning on quality of life in patients with psychogenic nonepileptic seizures versus epilepsy. Epilepsia. 2011 Feb;52(2):292-300. doi: 10.1111/j.1528-1167.2010.02765.x. Epub 2011 Feb 7. PMID 21299547
- [Result] LaFrance WC Jr, Baird GL, Barry JJ, Blum AS, Frank Webb A, Keitner GI, Machan JT, Miller I, Szaflarski JP; NES Treatment Trial (NEST-T) Consortium. Multicenter pilot treatment trial for psychogenic nonepileptic seizures: a randomized clinical trial. JAMA Psychiatry. 2014 Sep;71(9):997-1005. doi: 10.1001/jamapsychiatry.2014.817. PMID 24989152